CLINICAL TRIAL: NCT06951789
Title: Effect of Molecular Hydrogen Inhalation on Metabolic Response in Healthy Females During Low-intensity Exercise on a Bicycle Ergometer: A Randomized, Double-blind, Placebo-controlled Crossover Trial
Brief Title: Effect of Molecular Hydrogen Inhalation on Metabolic Response During Low-intensity Exercise on a Bicycle Ergometer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Assistant professor, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FTK_2024_101
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Respiratory Quotient Measurement
MeSH Terms: interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular hydrogen (Experimental): Molecular hydrogen inhalation for 20 min at rest and 30 min during exercise.
  Interventions: Other: Molecular hydrogen
- Placebo (Placebo Comparator): Placebo inhalation for 20 min at rest and 30 min during exercise.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Molecular hydrogen — Hydrogen gas, purity >99.9%, flow rate 600 ml/min (two generators 300 ml/min each).
  Other Names: i300 Hydrogen Generator, H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Molecular hydrogen
Other: Placebo — Ambient air, flow rate 600 ml/min (two pumps 300 ml/min each).
  Other Names: i300 Hydrogen Generator (placebo), H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Placebo

SUMMARY:
This trial evaluates the effect of molecular hydrogen inhalation on metabolic response, heart rate, and rating of perceived exertion in healthy females during 30 minutes of exercise on a bicycle ergometer.

DETAILED DESCRIPTION:
The objective of this randomized, double-blind, placebo-controlled crossover trial is to assess the effect of molecular hydrogen inhalation on metabolic response during 20 min of rest and during exercise on a bicycle ergometer with a workload of 0.5 W/kg for 10 min, 0.75 W/kg for 10 min, and 1 W/kg for 10 min. The trial recruits healthy females aged 20-35 years and the planned sample size is 20. The trial consists of two experimental sessions, one using molecular hydrogen inhalation and the other using placebo inhalation. The washout period between sessions is one week. Randomization of the order of the sessions is performed using a computer random generator. Molecular hydrogen is produced using a hydrogen generator via electrolysis of water and administered through a mouthpiece. Ambient air is used for placebo inhalation. Molecular hydrogen is colorless, odorless, and tasteless, making it indistinguishable from placebo by the human senses. During the session, the following variables are measured: ventilation, oxygen uptake, respiratory exchange ratio, heart rate, rating of perceived exertion, and oxygen saturation. Energy expenditure, fat oxidation rate and carbohydrates oxidation rate are calculated from oxygen uptake and respiratory exchange ratio. Statistical analysis is performed at the 0.05 significance level and data are evaluated using analysis of variance for repeated measures with Fisher's post hoc tests.

ELIGIBILITY:
Inclusion Criteria:

* Free of major diseases.
* Signed informed consent.

Exclusion Criteria:

* Acute conditions contraindicating laboratory testing of exercise.
* Cardiorespiratory disease.
* Pharmacotherapy affecting metabolism.
* Musculoskeletal problems.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Respiratory exchange ratio | Change after 1 week of crossover.
  Respiratory exchange ratio is measured with Ergostik analyser (Geratherm Respiratory, Bad Kissinger, Germany) breath by breath during the session and averaged over 5 min windows for subsequent analysis.

SECONDARY OUTCOMES:
Ventilation | Change after 1 week of crossover.
  Ventilation is measured with Ergostik analyser (Geratherm Respiratory, Bad Kissinger, Germany) breath by breath during the session and averaged over 5 min windows for subsequent analysis.
Oxygen uptake | Change after 1 week of crossover.
  Oxygen uptake is measured with Ergostik analyser (Geratherm Respiratory, Bad Kissinger, Germany) breath by breath during the session and averaged over 5 min windows for subsequent analysis.
Heart rate | Change after 1 week of crossover.
  Heart rate is recorded by Polar H10 chest strap (Polar, Kempele, Finland) during the session and averaged over 5 min windows for subsequent analysis.
Rating of perceived exertion | Change after 1 week of crossover.
  Participants are asked to subjectively rate their perceived exertion at specified time points (at the end of rest, after 10, 20, and 30 min of exercise). The Borg's scale 6 (no exertion) and 20 (maximal exertion) is used.

OTHER OUTCOMES:
Oxygen saturation | Change after 1 week of crossover.
  Oxygen saturation is measured with pulse oximeter (Onyx Vantage 9590, Nonin Medical, Plymouth, MN) at specified time points (every 5 min at rest and every 2,5 min during exercise).

CONTACTS AND LOCATIONS:
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: Beginning 1 month after the publication of results with no end date.